CLINICAL TRIAL: NCT04853758
Title: Angiotensin Receptor-Neprilysin Inhibition in Chagas Cardiomyopathy With Reduced Ejection Fraction: Randomized Trial ANSWER-HF
Brief Title: Angiotensin Receptor-Neprilysin Inhibition in Chagas Cardiomyopathy With Reduced Ejection Fraction: ANSWER-HF.
Acronym: ANSWER-HF
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: InCor Heart Institute (Other)
Responsible Party: Principal Investigator, FELIX JOSÉ ALVAREZ RAMIRES, Principal Investigator, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 33360220500000068
Record Dates: First submitted 2021-04-06; First posted 2021-04-21 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Chagas Cardiomyopathy
Keywords: Heart Failure; Chagas Disease; Chagas Cardiomyopathy; Sacubitril/Valsartan
MeSH Terms: conditions — Chagas Cardiomyopathy; Heart Failure; Chagas Disease | interventions — sacubitril; Valsartan; sacubitril and valsartan sodium hydrate drug combination; Enalapril; Angiotensin-Converting Enzyme Inhibitors

STUDY DESIGN:
Intervention Model Description: The ANSWER-HF will be a clinical, randomized, single-center, prospective, double-blind, controlled study. It will include 200 consecutive participants. This study will evaluate the benefit of sacubitril/valsartan compared with enalapril in patients with HF due to Chagas cardiomyopathy, with reduced ejection fraction(EF). Inclusion criteria are a positive serology for Chagas; age > 18 years old; NYHA HF and functional class II, III or IV; LVEF <40% at least in the last 3 months; patients using a beta-blocker with stable dose (1 month) and optimized; and using ACEI or ARB with a stable dose (1 month) and optimized. Exclusion criteria are participants who do not agree to participate in the study or do not want to receive sacubitril/ valsartan; with symptomatic hypotension; with SBP lower than 95 mmHg on randomization; with ClCr less than 30 mL/min; potassium > 5.2 mmol/L; and with a history of angioedema or who experienced severe side effects with ACE inhibitors.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Randomization will be carried out by the Heart Institute - School of Medicine of the University of São Paulo (InCor), using a RedCap platform, with blinded randomization being performed 1:1 for each arm of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sacubitril/Valsartan (Active Comparator): 100 consecutive participants randomized independently at the Heart Institute - School of Medicine of the University of São Paulo (InCor),will receive sacubitril/valsartan.
  Interventions: Drug: Sacubitril / Valsartan Oral Tablet [Entresto]
- Enalapril (Active Comparator): 100 consecutive participants randomized independently at the Heart Institute - School of Medicine of the University of São Paulo (InCor),will receive enalapril.
  Interventions: Drug: Enalapril

INTERVENTIONS:
Drug: Sacubitril / Valsartan Oral Tablet [Entresto] — 100 consecutive participants randomized independently at the Heart Institute - School of Medicine of the University of São Paulo (InCor),will receive sacubitril/valsartan for 6 months.
  Other Names: Angiotensin receptor-neprilisin inhibitor (ARNI)
  Arms: Sacubitril/Valsartan
Drug: Enalapril — 100 consecutive participants randomized independently at the Heart Institute - School of Medicine of the University of São Paulo (InCor),will receive enalapril for 6 months.
  Other Names: Angiotensin converting enzyme inhibitors (ACE inhibitors)
  Arms: Enalapril

SUMMARY:
Chagas disease is considered by the World Health Organization (WHO) as one of the most neglected tropical diseases in the world, having relevance in many Latin America countries. In addition, it already affects North America, Europe, Asia and Oceania. Some studies suggest that chagasic heart failure has a worse prognosis, with up to 50% shorter survival than other etiologies. The PARADIGM-HF (Prospective Comparison of Angiotensin Receptor Blocker-Neprilysin Inhibitor With Angiotensin-Converting Enzyme Inhibitor to Determine Impact on Global Mortality and Morbidity in Heart Failure) study showed 20% reduction in mortality comparing sacubitril/valsartan with the standard treatment with ACE (angiotensin converting enzyme) inhibitors. In the scenario of chagasic cardiomyopathy, a post hoc analysis of PARADGIM-HF was reported on 113 patients. Reduced risk of cardiovascular death or hospitalization for HF was noted in the group treated with sacubitril/valsartan. Attention was drawn the study's limitations that included the small number of patients and reduced statistical power. Therefore, the benefit of this new class remains uncertain in heart failure due to Chagas cardiomyopathy. The ANSWER-HF Trial will be a clinical, randomized, single-center, prospective, double-blind, controlled study. It will include 200 consecutive participants with Chagas cardiomyopathy and left ventricular ejection fraction less than 40% randomized independently. The objective of this study is to evaluate the benefit of sacubitril/valsartan compared with enalapril in patients with heart failure due to Chagas cardiomyopathy, with reduced ejection fraction. The primary endpoint of the study is the change of left ventricular ejection fraction determined by transthoracic echocardiography. Secondary endpoints include: assessment of ventricular arrhythmias; evaluation of functional class; assessment of functional capacity; assessment of ventricular remodeling; and evaluation of biomarkers. The patients will be followed for 6 months after treatment start. All patients will be undergone to Doppler Echocardiography, 24-hour Holter, 6-minute walk test, Biochemical and hematological exams and Biomarkers at the baseline and after 6 months.

DETAILED DESCRIPTION:
Introduction: Chagas disease (CD) is an infectious parasitic disease caused by the protozoan Trypanosoma cruzi. It is considered by the World Health Organization (WHO) as one of the most neglected tropical diseases in the world, having relevance in many Latin America countries. In addition, it already affects North America, Europe, Asia and Oceania due to current migration patterns. In the chronic phase, about 70% of individuals have no symptoms and routine complementary examinations related to the heart and digestive system do not show any changes. The other 30% of patients can develop the cardiac and/or digestive form of which about 10% may progress to severe heart disease. Chagasic cardiomyopathy is associated with major heart failure, sudden death, often due to severe arrhythmias and thromboembolic phenomena. This cardiomyopathy has a higher degree of myocardial fibrosis compared with any other etiology. Furthermore, some studies suggest that chagasic heart failure has a worse prognosis, with up to 50% shorter survival than survival with other etiologies, such as ischemic disease and idiopathic dilated cardiomyopathy. The pharmacological treatment of heart failure in Chagas disease comprises neurohormone blockers as is the case for angiotensin II converting enzime (ACE) inhibitors, angiotensin II (AII) receptor blocker (ARBs), beta-blockers and mineralocorticoid antagonists. In 2014 with the publication of the PARADIGM-HF study, a new drug class (ARNI: angiotensin receptor-neprilisin inhibitor) was proposed showing a 20% reduction in mortality compared with the standard treatment with ACE inhibitors. Sacubitril/valsartan is the first molecule of this class. This new molecule acts by blocking AII AT1 (angiotensin type 1) receptors, and therefore, attenuating the harmful effects of this peptide. It also promotes the blocking of the degradation of natriuretic peptides, increasing the protective effects of this family of proteins. In the scenario of chagasic cardiomyopathy, a post hoc analysis of PARADGIM-HF was conducted by Ramires and colleagues who reported on 113 patients treated with sacubitril/valsartan or enalapril. Reduced risk of cardiovascular death or hospitalization for HF was noted in the group treated with sacubitril/valsartan. Attention was drawn the study's limitations that included the small number of patients and reduced statistical power. Therefore, the benefit of this new class remains uncertain in heart failure due to Chagas cardiomyopathy. Knowing that chagasic cardiomyopathy is characterized by intense myocardial fibrosis, inflammation and oxidative stress, and with sacubitril/valsartan being the molecule that has a protective effect in exactly these same mechanisms, our hypothesis is that this drug may improve myocardial remodeling, and therefore it may modulate ventricular function, arrhythmias and functional capacity.

Methods: The ANSWER-HF Trial will be a clinical, randomized, single-center, prospective, double-blind, controlled study. It will include 200 consecutive participants randomized independently. The objective of this study is to evaluate the benefit of sacubitril/valsartan compared with enalapril in patients with heart failure due to Chagas cardiomyopathy, with reduced ejection fraction. Endpoints: The primary endpoint of the study is the change of left ventricular ejection fraction (LVEF) determined by transthoracic echocardiography. Secondary endpoints include: assessment of ventricular arrhythmias; evaluation of functional class; assessment of functional capacity; assessment of ventricular remodeling; and evaluation of biomarkers. Security outcomes include systolic blood pressure (SBP) less than 95 mmHg; renal function assessed by GFR (glomerular filtration rate) less than 30 mL/min; serum potassium > 5.2 mmol/L; and angioedema; whereas, exploratory outcomes are hospitalization for heart failure and mortality from all causes. Randomization: Randomization will be carried out using a RedCap platform blinded randomization being performed 1:1 for each arm of the study. Treatment Procedure and Strategies: The selected patients will go through the first visit (selection - V0), when the inclusion and exclusion criteria will be evaluated. If these criteria are met, the informed consent form (ICF) will then be presented and clarified. After all doubts are resolved, the patient or his or her legal representative must sign it. In this selection visit, the baseline tests that make up the inclusion/exclusion criteria (biochemical profile and echocardiogram) will be requested. Two weeks later, on visit 1 (randomization - V1), the tests performed will be analyzed and, if the patients' eligibility is confirmed, the patients will be randomized for each arm of the study. At this visit, baseline exams for the study (Holter, 6-minute walk test and pre-defined biomarkers) will be required. After two weeks, on visit 2 (V2) a new clinical evaluation will be carried out, and with no clinical exclusion criteria (pre-defined blood pressure levels and creatinine clearance), patients will receive the study medication. After two weeks, on visit 3 (V3), a new clinical evaluation will be carried out and the medication will be titrated according to that clinical evaluation. After 2 weeks, on visit 4 (V4), a new clinical evaluation and titration, if possible, will be conducted. After 4 weeks, on visit 5 (V5), a new clinical and biochemical assessment will be carried out, in addition to titration of the medication according to blood pressure levels. After 8 weeks on visit 6 (V6), clinical evaluation and medication titration will be performed according to blood pressure levels. Finally, after another 8 weeks, on visit 7 (V7), a new clinical and biochemical evaluation will be performed, in addition to a 6-minute walk test, transthoracic echocardiography, Holter and biomarker collection. Therefore, the study will be followed up for 6 months. Withdrawal and discontinuation: Despite the limited duration of the study, participants have the right to withdraw from the clinical investigation at any time and for any reason, without prejudice to their care. Doppler Echocardiography: All patients will undergo two-dimensional echocardiography with tissue Doppler, at the beginning and at the end of the protocol, under the guidelines of the cut and image plans published by the American Society of Echocardiography. Based on this guideline, the measurements of the left ventricular (LV) systolic and diastolic diameters will be quantified, as well as their respective volumes. The thickness of the LV interventricular septum and posterior wall will also be assessed and the LV ejection fraction will be quantified by the Simpsons method. The diastolic function will be measured using the transmitral Doppler obtaining the E (initial) and A (late) waves, E / A ratio and the E wave deceleration time (DT). The investigators will also obtain the tissue Doppler traces in the basal region of the septum and in the mitral lateral ring, to analyze the velocities of the s', e' and a' waves. 24-hour Holter: All patients in the study will undergo a 24-hour Holter monitoring, at the beginning and end of the protocol. The minimum, average and maximum heart rates will be analyzed, as well as the number, frequency and density of ventricular extrasystoles; episodes, duration and frequency of sustained or not sustained ventricular tachycardia; and finally the number and size of breaks. 6-minute walk test: The test will be applied according to the 2002 American Thoracic Society Guidelines. Before performing the test, patients will have a rest period of at least 10 minutes. During this period, data on blood pressure, pulse oximetry, dyspnea level (Borg scale), heart and respiratory rate should be evaluated, so that the test can begin. Biochemical and hematological exams: The laboratory tests evaluated in the study will be urea, creatinine, sodium, potassium, ionized calcium, magnesium, glycemia and C-reactive protein. These exams will be collected at V0, V5 and V7. Biomarkers: The NT-proBNP (N terminal-pro brain natriuretic peptide) will be evaluated. The concentrations of IL-6 (interleukin-6), TNFα (tumor necrosis factor alfa), Galectin-3 present in the patients' serum or plasma will be measured at the beginning and at the end of the protocol, through enzymatic immunoassays (ELISA) using specific company kits R & D Systems (Minneapolis, MN). For the analysis of microRNAs linked to inflammation and fibrosis, in the circulation, the investigators will follow the established protocol. The microRNAs selected for the study (mir-19a-3p; mir-30;mir-133 and housekeeping) synthesized by Applied Biosystems (Thermo Fisher Scientific Inc, USA) and their respective oligonucleotide sequences. Statistical Analysis: For the calculation of the sample size a few randomized studies have been conducted specifically in patients with Chagas cardiomyopathy. Most studies on heart failure do not distinguish the etiology of the disease, and therefore, all estimates assumed here consider that the expected effect based on the current literature is reflected in a similar way for chagasic patients. The PROVE-HF study (Januzzi et al., 2019) suggests that the improvement in EF in patients who receive sacubitril-valsartan is 5.2% with 95% CI (confidence interval) [4.8-5.6] at 6 months, which indicates a standard deviation of approximately 5.5% for this difference. The SOLVD (Studies of Left Ventricular Dysfunction) study (Kornstam et al., 1993) compared enalapril with placebo and showed an average improvement in EF of 3.0% in 1 year for patients in the enalapril group, with standard deviations at baseline and in 1 year similar to 5.5% from the previous study, which indicates that a standard deviation for the difference of 5.5% is also reasonable for the enalapril group. In addition, it is reasonable to assume that the effect in 6 months for the enalapril group is about half (1.5% or 2.0%), because PROVE-HF in one year had almost twice the effect (average improvement of 9.2%). In view of this, the investigators considers sample sizes for different scenarios, considering study powers of 80% and 90%, expected average differences between the improvements of the enalapril and sacubitril-valsartan groups varying from 2% to 5%, significance level of 5% for two-tailed hypotheses for a hypothesis test of comparison of proportions and 1:1 allocation (Chow et al., 2008). Because loss of follow-up (including death) is still possible, follow-up of these patients is a challenge. Including a 20% loss rate at the end of the estimate is suggested. Thus, the investigators could justify the study sample size of 182 (152 + ~ 20%) to identify an average difference of 2.5% of the improvement in EF with a standard deviation of 5.5%, considering a significance level of 5%, allocation 1:1, loss of follow-up of 20% and power of 80%. Statistical analysis: The normality of the quantitative variables will be assessed with the Shapiro-Wilks test. Parametric variables will be described as mean and standard deviation and compared using the Student t test. Nonparametric variables will be described with median and interquartile range and compared using the Mann-Whitney test. Categorical variables will be assessed using the chi-square test or Fisher exact test or likelihood ratio.Compliance Rules and Regulations: The protocol, the informed consent form and other documents related to the study was submitted to the Ethics Committee (CEP)/Institutional Review Board (CRI). The study will be carried out in accordance with the Declaration of Helsinki and Good Clinical Practice (GCP). Data storage and Quality Assurance and Management: It is expected that all data entered in REDCAP will have source documentation available. Data collection will be performed through an electronic case report form (eCRF).

ELIGIBILITY:
Inclusion Criteria:

1. Positive serology for Chagas;
2. Age > 18 years old;
3. New York Heart Association (NYHA) heart failure and functional class II, III or IV;
4. Left ventricular ejection fraction <40% at least in the last 3 months;
5. Patients using a beta-blocker with stable dose (last 4 weeks) and optimized;
6. Patients using ACEI or ARB with a stable dose (last 4 weeks) and optimized.

Exclusion Criteria:

1. Participants who do not agree to participate in the study
2. Participants who do not want to receive sacubitril/ valsartan medication;
3. Patients with symptomatic hypotension;
4. Patients with systolic blood pressure (SBP) lower than 95 mmHg on randomization;
5. Patients with creatinine clearance (ClCr) less than 30 mL/min;
6. Patients with serum potassium > 5.2 mmol/L;
7. Patients with a history of angioedema or who experienced severe side effects with ACE inhibitors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-05-06 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Change of left ventricular ejection fraction (LVEF) | 6 months
  The primary endpoint of the study will be studied by transthoracic echocardiography. The LVEF will be evaluated using Simpson method.
Win Ratio Analysis | 6 meses
  Hierarchical composite analysis composed of: 1. Time to cardiovascular death; 2. Time to first heart failure hospitalization; 3. Relative change in NT-proBNP from baseline to final visit; 4. Relative change in left ventricular ejection fraction from baseline to final visit

SECONDARY OUTCOMES:
Number of premature ventricular beats | 6 months
  It will be measured by 24 hour Holter counting the absolute number of premature ventricular beats.
Percentage of premature ventricular beats. | 6 months
  It will be measured by 24 hour Holter counting the percentage of premature ventricular beats.
Ventricular arrhythmias density | 6 months
  It will be measured by 24 hour Holter counting the non-sustained ventricular tachycardia rates.
Sustained ventricular tachycardia rates | 6 months
  It will be measured by 24 hour Holter counting the sustained ventricular tachycardia rates.
New York Heart Association functional class | 6 months
  This variable will be clinically evaluate during visits and will be analyzed in 6 months.
Ventricular remodeling - left ventricular systolic diameter | 6 months
  It will be measured by echocardiography and the variable studied will be left ventricular systolic diameter
Ventricular remodeling - left ventricular diastolic diameter. | 6 months
  It will be measured by echocardiography and the variable studied will be left ventricular diastolic diameter.
Ventricular remodeling - left ventricular systolic volume. | 6 months
  It will be measured by echocardiography and the variable studied will be left ventricular systolic volume.
Ventricular remodeling - left ventricular diastolic volume | 6 months
  It will be measured by echocardiography and the variable studied will be left ventricular diastolic volume.
Ventricular remodeling - thickness of the interventricular septum. | 6 months
  It will be measured by echocardiography and the variable studied will be thickness of the interventricular septum.
Ventricular remodeling - thickness of the left ventricular posterior wall.. | 6 months
  It will be measured by echocardiography and the variable studied will be thickness of the LV posterior wall.
Safety biochemical biomarkers - urea. | 3 and 6 months
  This evaluation will analyse blood urea (mg/dL).
Safety biochemical biomarkers - creatinine. | 3 and 6 months
  This evaluation will analyse blood creatinine (mg/dL).
Evaluation of biomarkers - systemic cytokines. | 6 months
  This evaluation will be measured using ELISA for systemic cytokines (IL-6, TNF, Galectin-3) pg/ml
Evaluation of biomarkers - MicroRNA. | 6 months
  This evaluation will be measured using molecular biology for systemic expression for MicroRNA (MIR133, MIR19a,MIR30a)
Evaluation of biomarkers - NT-proBNP | 6 months
  This evaluation will be measured analysing NT-proBNP (pg/ml)
Safety biochemical biomarkers - potassium. | 3 and 6 months
  This evaluation will analyse blood potassium (mEq/L).
Safety biochemical biomarkers - sodium. | 3 and 6 months
  This evaluation will analyse blood sodium (mEq/L).

CONTACTS AND LOCATIONS:
Overall Officials: Felix José JA Ramires, MD,PhD, Principal Investigator — Instituto do Coração - INCORHCFMUSP
Locations (1):
- Heart Institute (Incor) University of Sao Paulo, São Paulo, Brazil

REFERENCES:
- [Result] Hotez PJ, Fenwick A, Savioli L, Molyneux DH. Rescuing the bottom billion through control of neglected tropical diseases. Lancet. 2009 May 2;373(9674):1570-5. doi: 10.1016/S0140-6736(09)60233-6. No abstract available. PMID 19410718
- [Result] Bocchi EA, Rassi S, Guimaraes GV; Argentina, Chile, and Brazil SHIFT Investigators. Safety profile and efficacy of ivabradine in heart failure due to Chagas heart disease: a post hoc analysis of the SHIFT trial. ESC Heart Fail. 2018 Jun;5(3):249-256. doi: 10.1002/ehf2.12240. Epub 2017 Dec 20. PMID 29266804
- [Result] Ianni BM, Arteaga E, Frimm CC, Pereira Barretto AC, Mady C. Chagas' heart disease: evolutive evaluation of electrocardiographic and echocardiographic parameters in patients with the indeterminate form. Arq Bras Cardiol. 2001 Jul;77(1):59-62. doi: 10.1590/s0066-782x2001000700006. PMID 11500748
- [Result] Araujo FG, Chiari E, Dias JC. Demonstration of Trypanosoma cruzi antigen in serum from patients with Chagas' disease. Lancet. 1981 Jan 31;1(8214):246-9. doi: 10.1016/s0140-6736(81)92088-2. PMID 6109902
- [Result] Carod-Artal FJ, Gascon J. Chagas disease and stroke. Lancet Neurol. 2010 May;9(5):533-42. doi: 10.1016/S1474-4422(10)70042-9. PMID 20398860
- [Result] Barretto AC, Higuchi ML, da Luz PL, Lopes EA, Bellotti G, Mady C, Stolf N, Arteaga-Fernandez E, Pileggi F. [Comparison of histologic changes in Chagas' cardiomyopathy and dilated cardiomyopathy]. Arq Bras Cardiol. 1989 Feb;52(2):79-83. Portuguese. PMID 2596992
- [Result] Mady C, Cardoso RH, Barretto AC, da Luz PL, Bellotti G, Pileggi F. Survival and predictors of survival in patients with congestive heart failure due to Chagas' cardiomyopathy. Circulation. 1994 Dec;90(6):3098-102. doi: 10.1161/01.cir.90.6.3098. PMID 7994859
- [Result] Shen L, Ramires F, Martinez F, Bodanese LC, Echeverria LE, Gomez EA, Abraham WT, Dickstein K, Kober L, Packer M, Rouleau JL, Solomon SD, Swedberg K, Zile MR, Jhund PS, Gimpelewicz CR, McMurray JJV; PARADIGM-HF and ATMOSPHERE Investigators and Committees. Contemporary Characteristics and Outcomes in Chagasic Heart Failure Compared With Other Nonischemic and Ischemic Cardiomyopathy. Circ Heart Fail. 2017 Nov;10(11):e004361. doi: 10.1161/CIRCHEARTFAILURE.117.004361. PMID 29141857
- [Result] McMurray JJ, Packer M, Desai AS, Gong J, Lefkowitz MP, Rizkala AR, Rouleau JL, Shi VC, Solomon SD, Swedberg K, Zile MR; PARADIGM-HF Investigators and Committees. Angiotensin-neprilysin inhibition versus enalapril in heart failure. N Engl J Med. 2014 Sep 11;371(11):993-1004. doi: 10.1056/NEJMoa1409077. Epub 2014 Aug 30. PMID 25176015
- [Result] Ramires FJA, Martinez F, Gomez EA, Demacq C, Gimpelewicz CR, Rouleau JL, Solomon SD, Swedberg K, Zile MR, Packer M, McMurray JJV. Post hoc analyses of SHIFT and PARADIGM-HF highlight the importance of chronic Chagas' cardiomyopathy Comment on: "Safety profile and efficacy of ivabradine in heart failure due to Chagas heart disease: a post hoc analysis of the SHIFT trial" by Bocchi et al. ESC Heart Fail. 2018 Dec;5(6):1069-1071. doi: 10.1002/ehf2.12355. Epub 2018 Oct 9. No abstract available. PMID 30298996
- [Derived] Madrini V Jr, Souza PVR, Fernandes F, Ianni BM, Martins AS, Luzuriaga GJ, Fonseca KCB, Ribeiro ODN, da Cruz AB, Oliveira R, Antunes TL, Pessoa FG, Damiani LP, Quaglio LS, Correia VM, Antunes MO, Mady C, Guimaraes PO, Tavares CAM, Biselli B, Gruppi CJ, Mathias W Jr, Bihan DCSL, Bocchi EA, Lopes RD, Alvarez Ramires FJ; ANSWER-HF Investigators. Sacubitril-Valsartan vs Enalapril in Heart Failure Due to Chagas Disease: Primary Results of ANSWER-HF Randomized Trial. J Am Coll Cardiol. 2025 Nov 9:S0735-1097(25)10064-8. doi: 10.1016/j.jacc.2025.10.053. Online ahead of print. PMID 41396086
- See also: Sustaining the drive to overcome the global impact of neglected tropical diseases. Second WHO report on neglected tropical diseases — https://www.paho.org/fr/node/64408